CLINICAL TRIAL: NCT00932906
Title: Comparison of Four Different AED Training Methods in Three Different Age Groups
Brief Title: Comparison of Different Automated External Defibrillation (AED) Training Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Doczero (Other)
Collaborators: Laerdal Medical (Industry)
Responsible Party: Wiebe de Vries, Doczero
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Ed-2008-06
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Improvement of BLS/AED Training Programmes
Keywords: Education; Retention; Retrieval; Self training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- Instructor based training; <21 years (Placebo Comparator): The instructor based training is a 1.25 hour training as described by the ERC in their standard training program [ref; navragen bij Koen] and using the ERC PowerPoint presentation. There is one manikin and one AED trainer per six students. The group consists out of 12 students maximal, with one instructor per six students.
  Interventions: Other: Standard training
- Instructor based training; 21-50 years (Placebo Comparator): The instructor based training is a 1.25 hour training as described by the ERC in their standard training program [ref; navragen bij Koen] and using the ERC PowerPoint presentation. There is one manikin and one AED trainer per six students. The group consists out of 12 students maximal, with one instructor per six students.
  Interventions: Other: Standard training
- Instructor based training; >50 years (Placebo Comparator): The instructor based training is a 1.25 hour training as described by the ERC in their standard training program [ref; navragen bij Koen] and using the ERC PowerPoint presentation. There is one manikin and one AED trainer per six students. The group consists out of 12 students maximal, with one instructor per six students.
  Interventions: Other: Standard training
- Video Skill Training; <21 years (Experimental): Participants practise AED skills, watching a 4.5-min video in a single uninterrupted session. There is no instructor available. The video demonstrates the use of an AED; when to use it, how to turn it on, how to attach the electrodes, keeping distance and delivering a shock.
  Interventions: Other: Different self-training methods
- Video Skill Training; 21-50 years (Experimental): Participants practise AED skills, watching a 4.5-min video in a single uninterrupted session. There is no instructor available. The video demonstrates the use of an AED; when to use it, how to turn it on, how to attach the electrodes, keeping distance and delivering a shock.
  Interventions: Other: Different self-training methods
- Video Skill Training; >50 years (Experimental): Participants practise AED skills, watching a 4.5-min video in a single uninterrupted session. There is no instructor available. The video demonstrates the use of an AED; when to use it, how to turn it on, how to attach the electrodes, keeping distance and delivering a shock.
  Interventions: Other: Different self-training methods
- Video scenario training; <21 years (Experimental): Participants practises AED skills, watching a 9-min video in a single uninterrupted session. There is no instructor available. The video demonstrates the use of an AED; when to use it, how to turn it on, how to attach the electrodes, keeping distance and delivering a shock, and additional two scenarios, in each of which they practice the BLS/AED procedure.
  Interventions: Other: Different self-training methods
- Video scenario training; 21-50 years (Experimental): Participants practises AED skills, watching a 9-min video in a single uninterrupted session. There is no instructor available. The video demonstrates the use of an AED; when to use it, how to turn it on, how to attach the electrodes, keeping distance and delivering a shock, and additional two scenarios, in each of which they practice the BLS/AED procedure.
  Interventions: Other: Different self-training methods
- Video scenario training; >50 years (Experimental): Participants practises AED skills, watching a 9-min video in a single uninterrupted session. There is no instructor available. The video demonstrates the use of an AED; when to use it, how to turn it on, how to attach the electrodes, keeping distance and delivering a shock, and additional two scenarios, in each of which they practice the BLS/AED procedure.
  Interventions: Other: Different self-training methods
- Video demonstration training; <21 years (Experimental): Participants watch a 2.5 minutes video demonstration of the use of an AED, in a single uninterrupted session, without hands-on practice.
  Interventions: Other: Different self-training methods
- Video demonstration training; 21-50 years (Experimental): Participants watch a 2.5 minutes video demonstration of the use of an AED, in a single uninterrupted session, without hands-on practice.
  Interventions: Other: Different self-training methods
- Video demonstration training; >50 years (Experimental): Participants watch a 2.5 minutes video demonstration of the use of an AED, in a single uninterrupted session, without hands-on practice.
  Interventions: Other: Different self-training methods

INTERVENTIONS:
Other: Different self-training methods — Self training with MiniAnne Training Kit
  Arms: Video Skill Training; 21-50 years; Video Skill Training; <21 years; Video Skill Training; >50 years; Video demonstration training; 21-50 years; Video demonstration training; <21 years; Video demonstration training; >50 years; Video scenario training; 21-50 years; Video scenario training; <21 years; Video scenario training; >50 years
Other: Standard training — Instructor-based training meeting ERC directions
  Arms: Instructor based training; 21-50 years; Instructor based training; <21 years; Instructor based training; >50 years

SUMMARY:
This study is a prospective, randomized trial that compares the effectiveness and retention of four different training methods for the use of an AED:

A. Traditional instructor based learning;

B. The use of a personal manikin with a DVD training to practice the necessary AED skills;

C. The use of a personal manikin with a DVD training to practice the necessary AED skills and additional scenario training;

D. Watching a 2.5 minutes DVD which shows the use of an AED.

It is hypnotised that there are no differences between these training methods, in which case method D is most efficient to reach large number of people to learn BLS/AED skills.

There are two interesting target groups to reach:

1. Younger people, as they might give the highest interest after training, as they normally live longer.
2. Older people as they are member of the most important group in risk and have therefore a higher change of being a witness of cardiac arrest.

As there might be differences in the results between different training methods than can be related to age, each training group is distinguished to three different groups:

1. 21 years of younger;
2. between 21 and 50 years;
3. older than 50 years.

It is hypnotised that there are no differences between younger and older students within each of the four training methods.

ELIGIBILITY:
Inclusion Criteria:

* willing to follow a BLS/AED course up to 2h

Exclusion Criteria:

* CPR training within the last five years
* professional health care provider

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-06 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Kruskal-Wallis test | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wiebe de Vries, MSc, Principal Investigator — Doczero; Koenraad Monsieurs, Professor, Study Director — University Hospital, Ghent; Joost Bierens, Professor, Study Chair — VU Medical Centre; Rudolph Koster, PhD MD, Study Chair — Academical Medical Centre Amsterdam; Nigel M Turner, PhD MD, Study Chair — Medicine, Wilhelmina Children Hospital - University Medical Centre Utrecht